CLINICAL TRIAL: NCT04910100
Title: Randomized, Multicenter, Observer-Masked Study to Compare Safety/Efficacy of Nebivolol Suspension 0.5% or 1.0%, or Timolol Suspension 0.5% to Timolol Solution 0.5% in Participants With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: Nebivolol 0.5, 1.0, or Timolol 0.5 Suspension Compared to Timolol 0.5 Solution to Treat Glaucoma/Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Betaliq, Inc. (Industry)
Collaborators: Trial Runners, LLC (Other); Summit Analytical LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTQ-1901-1902-201
Record Dates: First submitted 2021-05-10; First posted 2021-06-02 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized in a 1:1:1:1 ratio to 4 treatment arms: nebivolol 0.5% ophthalmic suspension; nebivolol 1.0% ophthalmic suspension; timolol 0.5% ophthalmic suspension; and timolol 0.5% ophthalmic solution.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is observer masked. The study medication will be provided in foil pouches contained in identical-appearing boxes. An unmasked staff member not involved in performing study endpoint-related procedures (i.e., IOP measurement) will be responsible for providing dosing instructions, dispensing study medication, and conducting study medication accountability and dosing compliance assessment. The identity of the study medications will be masked to the Investigator and study personnel responsible for study endpoint-related procedures. IOP measurements will be performed by the Investigator/designee who will be masked to the readout of the tonometer, which will be read and entered into the source documentation (whether electronic or paper) by a second staff member once the Investigator/designee reaches the correct applanation effect in the slit lamp.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nebivolol Ophthalmic Suspension 1 Percent (Experimental): Administered twice daily to both eyes for 84 days (12 weeks)
  Interventions: Drug: Nebivolol Ophthalmic Suspension 1 Percent
- Nebivolol Ophthalmic Suspension 0.5 Percent (Experimental): Administered twice daily to both eyes for 84 days (12 weeks)
  Interventions: Drug: Nebivolol Ophthalmic Suspension 0.5 Percent
- Timolol Ophthalmic Suspension 0.5 Percent (Experimental): Administered twice daily to both eyes for 84 days (12 weeks)
  Interventions: Drug: Timolol Ophthalmic Suspension 0.5 Percent
- Timolol Ophthalmic Solution 0.5 Percent (Active Comparator): Administered twice daily to both eyes for 84 days (12 weeks)
  Interventions: Drug: Timolol Ophthalmic Solution 0.5 Percent

INTERVENTIONS:
Drug: Nebivolol Ophthalmic Suspension 1 Percent — 1 drop instilled into each eye twice daily
  Arms: Nebivolol Ophthalmic Suspension 1 Percent
Drug: Nebivolol Ophthalmic Suspension 0.5 Percent — 1 drop instilled into each eye twice daily
  Arms: Nebivolol Ophthalmic Suspension 0.5 Percent
Drug: Timolol Ophthalmic Suspension 0.5 Percent — 1 drop instilled into each eye twice daily
  Arms: Timolol Ophthalmic Suspension 0.5 Percent
Drug: Timolol Ophthalmic Solution 0.5 Percent — 1 drop instilled into each eye twice daily
  Arms: Timolol Ophthalmic Solution 0.5 Percent

SUMMARY:
The purpose of this study is to evaluate the safety (in the eye and throughout the body) and effectiveness of nebivolol (0.5 and 1 percent) and timolol (0.5 percent) eye drop suspensions. These eye drops will be compared to timolol 0.5 percent eye drop solution in participants with open angle glaucoma (the most common type of glaucoma) or high eye pressure (ocular hypertension).

DETAILED DESCRIPTION:
The study will enroll 240 participants (60 in each treatment arm) who will be treated for 84 days (12 weeks). Participants will have OAG (open angle glaucoma) or OHT (ocular hypertension) in both eyes (OAG in one eye and OHT in the follow eye is acceptable) that requires therapy and elevated IOP (intraocular pressure) adequately controlled on no more than 2 ocular hypertensive medications. Participants with OHT on no ocular hypotensive medications are acceptable. After being informed about the study and potential risks, participants giving written informed consent will undergo an washout period, if required, from previous glaucoma medications (28 days for prostaglandin analogs, rho-associated protein kinase inhibitors, or beta blockers; 14 days for adrenergic agonists; and 5 days for muscarinic agonists or carbonic anhydrase inhibitors). Eligible participants must have unmedicated IOP measurements at Visit 3/Baseline ≥ 22 and ≤ 34 mm Hg at 8:00 AM and ≥ 18 and ≤ 34 mm Hg at 10:00 AM and 4:00 PM (each qualifying eye must fall within the required IOP range at all 3 time points and must be at least 22 mm Hg at each consecutive measurement at the 8:00 AM time point). Both eyes will be treated twice daily. Study visits will comprise Visit 1/Screening/Day -35 to -1, Visit 2/Washout Safety Check/Day -14 ± 3 (performed for participants undergoing 28-day washout periods at the Investigator's discretion), Visit 3/Qualification/Baseline/Day 1, Visit 4/Day 15 ± 3, Visit 5/Day 42 ± 3, and Visit 6/Day 84 ± 3. At Visits 4, 5, and 6, participants will be evaluated at 8:00 AM, at 2 hours after study medication dosing at the clinical site (approximately 10:00 AM), and at 4:00 PM (each ± 30 minutes). All ophthalmic assessments will be performed bilaterally.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and sign an informed consent form prior to any study related procedures.
2. Able to administer or have a caregiver accurately administer an eye drop.
3. Have POAG or OHT in both eyes that requires therapy for IOP and is adequately controlled, in the opinion of the Investigator, on no more than 2 ocular hypotensive medications (fixed dose combinations count as 2 medications). Subjects with OHT on no ocular hypotensive medication are acceptable. Presence of POAG in one eye and OHT in the fellow eye is acceptable.

3. Able, in the opinion of the Investigator, to safely discontinue use of ocular hypotensive medications, if applicable, and undergo the appropriate required washout period for ocular hypotensive medications prior to Visit 3/Qualification/Baseline.

4. At Visit 3/Qualification/Baseline, at least one eye must have unmedicated (post washout) IOP ≥ 22 and ≤ 34 mm Hg at 8:00 AM and ≥ 18 and ≤ 34 mm Hg at 10:00 AM and 4:00 PM in the same eye(s) qualifying at the Visit 3 8:00 AM time point. The IOP must be at least 22 mm Hg at each consecutive measurement at the 8:00 AM time point.

5. No significant VF (visual field) loss, defined as a mean deviation in either eye greater than - 12 dB or a central point of fixation < 5 dB in either eye. If the VF performed at or within 90 days prior to Visit 1 does not meet study required parameters, it may be repeated (test should be prior to randomization at Visit 3/Qualification/Baseline).

6. Best corrected visual acuity (BCVA) of +0.6 logMAR or better in both eyes at Visit 1/Screening and Visit 3/Qualification/Baseline.

7. Central corneal thickness ≥ 480 and ≤ 600 μm in both eyes. Pachymetry within 90 days prior to Screening is acceptable.

8. Shaffer gonioscopic grade ≥ 3 (in at least 3 quadrants) in both eyes. Gonioscopy within 90 days prior to randomization is acceptable.

9. Female subjects must be 1-year postmenopausal, surgically sterilized (total hysterectomy, bilateral oophorectomy or bilateral tubal ligation > 90 days prior to Visit 1/Screening), or women of childbearing potential with a negative urine pregnancy test at Visit 1/Screening and Visit 3/Qualification/Baseline who are not breastfeeding or planning a pregnancy during the study. Women of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include the use of at least one of the following:

* Intrauterine (IUD) device
* Hormonal contraceptive (oral, injection, patch, implant, ring); subjects must have been on the same hormonal contraceptive for ≥ 90 days prior to Visit 1/Screening
* Double barrier method (spermicide used with either a condom or diaphragm)
* Abstinence

Exclusion Criteria:

Ocular

1. Intraocular pressure ˃ 34 mm Hg in either eye at Visit 1/Screening, Visit 2/Washout Safety Check, or Visit 3/Qualification/Baseline.
2. Other forms of glaucoma in either eye, e.g., congenital glaucoma, closed-angle glaucoma, uveitic glaucoma, pseudoexfoliation or pigment dispersion syndrome, or history of angle closure. Narrow angles treated with peripheral iridotomy are allowed if at least 4 months status post iridotomy.
3. Current or recent (within 30 days prior to Visit 1/Screening) clinically significant ocular infection or inflammation, in the opinion of the Investigator, in either eye.
4. History of conjunctivitis within 90 days prior to Visit 1/Screening, or history of herpes simplex or herpes zoster in either eye.
5. Clinically significant ocular disease, in the opinion of the Investigator, in either eye (including, but not limited to corneal edema, uveitis, severe dry eye, proliferative diabetic retinopathy or macular degeneration) that might interfere with the study, confound study results, or put the subject at increased risk.
6. Have a cup-to disc (CD) ratio > 0.8 at Visit 1/Screening in either eye.
7. Intravitreal steroid injections within 6 months prior to Visit 1/Screening. Subconjunctival or subtenon steroid injections within 90 days prior to Visit 1/Screening.
8. Use of topical ocular medications within 30 days prior to Visit 1/Screening other than ocular hypotensive medications and medications used as part of an eye examination. Artificial tears may be used during this period provided the use is not required for severe dry eye disease.
9. Clinically significant ocular trauma or incisional ocular surgery (including routine cataract surgery) in either eye within 6 months prior to Visit 1/Screening. Glaucoma filtering surgery, or minimally invasive glaucoma surgery within 12 months prior to Visit 1/Screening. Laser surgery for IOP reduction within 6 months prior to Visit 1/Screening. Non-incisional ocular surgery or non-glaucomatous laser treatment within 90 days prior to Visit 1/Screening.
10. Refractive surgery in either eye (i.e., radial keratotomy, photorefractive keratectomy [PRK], laser-assisted in situ keratomileusis [LASIK], corneal cross-linking, limbal relaxing incision) within 6 months prior to Visit 1/Screening.
11. Any ocular (e.g., corneal) abnormality preventing accurate assessment of IOP.
12. Contact lens wear within 1 week prior to Visit 1/Screening or unwillingness to discontinue wear of contacts lenses prior to and during the study period.
13. Aphakia.

    General
14. Pregnancy or lactation.
15. Known hypersensitivity or contraindication to β-blockers (i.e., chronic obstructive pulmonary disease, bronchial asthma, unstable or abnormally low blood pressure or heart rate, second or third degree heart block or congestive heart failure, severe or unstable diabetes mellitus) that in the opinion of the Investigator may put the subject at risk from a topical ocular beta-blocker.
16. Have a condition or be in a situation which, in the Investigator's opinion, may put the subject at significant risk, confound study results, or interfere with the subject's participation in the study.
17. Clinically significant systemic disease (myasthenia gravis, hepatic, renal, endocrine, or cardiovascular disorders) that in the opinion of the Investigator might interfere with the study.
18. Use of systemic beta-adrenergic antagonists unless the dosage has been stable for 1 month prior to Visit 1/Screening and is expected to remain stable through the study period.
19. Use of systemic (oral, injectable, inhaled) or topical steroids within 30 days prior to Visit 1/Screening; topical dermatologic or intranasal steroids are acceptable provided the usage meets the criteria outlined in the Summary of Prohibited Medications and Procedures in the protocol.
20. Contraindication to the use of timolol, nebivolol, or any of the components of the investigational products.
21. Changes to systemic medication that could have an effect on IOP within 28 days prior to Visit 3/Qualification/Baseline.
22. Participation in any study of an investigational product within 30 days prior to Visit 1/Screening.
23. History of substance abuse within 1 year prior to Visit 1/Screening.
24. Screening and enrollment of employees or relatives of employees of the clinical site.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Peterson, Study Director — Trial Runners, LLC
Locations (1):
- Site 0012, Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 226 subjects were recruited and treated at 19 clinical investigation sites over a 12 month period commencing on 15 April 2021 and completing on 31 March 2022
Pre-assignment Details: Following successful completion of screening based on protocol specified inclusion and exclusion criteria and a wash out period of up to 28 days subjects were treated with investigational medication twice daily for 84 days.
Period: Overall Study
Arm/Group | Nebivolol Ophthalmic Suspension 1 Percent | Nebivolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Solution 0.5 Percent
Started | 54 | 58 | 56 | 58
Completed | 49 | 51 | 55 | 54
Not Completed | 5 | 7 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol Ophthalmic Suspension 1 Percent | Nebivolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Solution 0.5 Percent | Total
Number analyzed (Participants) | 54 | 58 | 56 | 58 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (13.92) | 67.6 (10.38) | 65.6 (12.71) | 66.0 (11.6) | 66.0 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 35 | 32 | 137
  Male | 18 | 24 | 21 | 26 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 11 | 11 | 43
  Not Hispanic or Latino | 43 | 48 | 45 | 47 | 183
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 20 | 18 | 20 | 74
  White | 37 | 38 | 37 | 37 | 149
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 58 | 56 | 58 | 226

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure Over 84 Days
Description: Measured utilizing a calibrated Goldmann tonometer; two consecutive IOP measurements of each eye will be performed. If the 2 measurements differ by more than 2 mm Hg, a third measurement will be taken. The primary efficacy analysis will be the between-group comparison of the mean IOP values in the study eye at 10AM, 2 hours postdose, and 4PM, at each of the Visit 4/Day 15, Visit 5/Day 42, and Visit 6/Day 84 visits (ie, a total of 9 between-group comparisons). A hierarchical analysis will be conducted to compare each of the investigational products against the comparator, timolol 0.5% ophthalmic solution, as follows: (1) nebivolol 1% ophthalmic suspension, (2) nebivolol 0.5% ophthalmic suspension, and (3) timolol ophthalmic suspension.
Time Frame: Over 84 days
Population: The analysis is performed at 9 different time points and compared to baseline (Visit 3 - Day 1), hence, the numbers analyzed at each time point differs from the overall number due to drop outs
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Nebivolol Ophthalmic Suspension 1 Percent | Nebivolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Solution 0.5 Percent
Number analyzed (Participants) | 52 | 56 | 55 | 57
mmHg
  Visit 4 - Day 15 - 8 am: number analyzed (Participants) | 51 | 56 | 55 | 57
  Visit 4 - Day 15 - 8 am | 22.0 [21.1 to 23.0] | 22.5 [21.6 to 23.4] | 18.8 [17.9 to 19.7] | 19.4 [18.5 to 20.3]
  Visit 4 - Day 15 - 10 am: number analyzed (Participants) | 51 | 54 | 55 | 57
  Visit 4 - Day 15 - 10 am | 20.4 [19.5 to 21.2] | 21.1 [20.3 to 21.9] | 17.7 [16.9 to 18.5] | 17.9 [17.1 to 18.8]
  Visit 4 - Day 15 - 4 pm: number analyzed (Participants) | 51 | 54 | 55 | 57
  Visit 4 - Day 15 - 4 pm | 19.8 [18.9 to 20.6] | 20.6 [19.8 to 21.4] | 18.2 [17.4 to 19.0] | 18.4 [17.6 to 19.2]
  Visit 5 - Day 42 - 8 am: number analyzed (Participants) | 50 | 52 | 55 | 55
  Visit 5 - Day 42 - 8 am | 21.8 [20.8 to 22.8] | 21.7 [20.7 to 22.7] | 19.0 [18.1 to 20.0] | 19.3 [18.4 to 20.3]
  Visit 5 - Day 42 - 10 am: number analyzed (Participants) | 49 | 51 | 55 | 55
  Visit 5 - Day 42 - 10 am | 20.2 [19.3 to 21.2] | 20.3 [19.4 to 21.3] | 17.8 [16.9 to 18.7] | 18.3 [17.4 to 19.2]
  Visit 5 - Day 42 - 4 pm: number analyzed (Participants) | 49 | 50 | 55 | 55
  Visit 5 - Day 42 - 4 pm | 20.1 [19.1 to 21.0] | 20.5 [19.5 to 21.5] | 18.4 [17.4 to 19.3] | 18.3 [17.4 to 19.2]
  Visit 6 - Day 84 - 8 am: number analyzed (Participants) | 48 | 49 | 54 | 54
  Visit 6 - Day 84 - 8 am | 21.2 [20.3 to 22.2] | 21.3 [20.4 to 22.2] | 18.5 [17.6 to 19.4] | 19.4 [18.6 to 20.3]
  Visit 6 - Day 84 -10 am: number analyzed (Participants) | 47 | 49 | 54 | 54
  Visit 6 - Day 84 -10 am | 20.1 [19.3 to 20.9] | 20.2 [19.4 to 21.0] | 17.9 [17.1 to 18.6] | 18.6 [17.8 to 19.3]
  Visit 6 - Day 84 - 4 pm: number analyzed (Participants) | 47 | 49 | 54 | 54
  Visit 6 - Day 84 - 4 pm | 19.8 [19.0 to 20.6] | 20.1 [19.3 to 20.8] | 18.1 [17.4 to 18.9] | 18.6 [17.9 to 19.4]
Statistical Analysis 1: Comparison: Timolol Ophthalmic Suspension 0.5 Percent vs Timolol Ophthalmic Solution 0.5 Percent; The primary efficacy analysis was the between group comparison of the mean IOP values in the study eye at each time point at each visit (a total of 9 between-group comparisons). A hierarchical analysis was conducted to compare each of the investigational products against the comparator, timolol 0.5% as follows: (1) Timolol Suspensions 0.5% (2) Nebivolol Suspension 1% (3) Nebivolol Suspension 0.5%; Test type: Non-Inferiority — To demonstrate noninferiority, the upper limits of the 2-sided 95% confidence interval for the difference between each comparison must be lower than 1.5 mmHg at all timepoints and lower than 1.0 mmHg for the majority of the timepoints (i.e. at least 5 of 9). This was a Phase 2 study and so the sample size was not based on a formal sample size calculation. The study was planned to provide sufficient data to power a Phase 3 study; Timepoints with Mean IOP < 1.5 mm Hg = 6
Statistical Analysis 2: Comparison: Timolol Ophthalmic Suspension 0.5 Percent vs Timolol Ophthalmic Solution 0.5 Percent; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Timepoints with Mean IOP < 1.0 mm Hg = 9
Statistical Analysis 3: Comparison: Nebivolol Ophthalmic Suspension 1 Percent vs Timolol Ophthalmic Solution 0.5 Percent; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Timepoints with Mean IOP < 1.5 mm Hg = 0
Statistical Analysis 4: Comparison: Nebivolol Ophthalmic Suspension 1 Percent vs Timolol Ophthalmic Solution 0.5 Percent; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Timepoints with Mean IOP < 1.0 mm Hg = 0
Statistical Analysis 5: Comparison: Nebivolol Ophthalmic Suspension 0.5 Percent vs Timolol Ophthalmic Solution 0.5 Percent; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Timepoints with Mean IOP < 1.5 mm Hg = 0
Statistical Analysis 6: Comparison: Nebivolol Ophthalmic Suspension 0.5 Percent vs Timolol Ophthalmic Solution 0.5 Percent; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Timepoints with Mean IOP < 1.0 mm Hg = 0

2. Secondary Outcome: Intraocular Pressure: Change From Baseline in Diurnal IOP at Each Visit
Description: Change from baseline (Visit 3/Qualification/Baseline) in the average of the 3 daily IOP measurements at Day 15, Day 42, and Day 84
Time Frame: Day 15: 8 AM ± 30 minutes, 2 hours post-dose ± 30 minutes, 4 PM ± 30 minutes; Day 42: 8 AM ± 30 minutes, 2 hours post-dose ± 30 minutes, 4 PM ± 30 minutes; Day 84: 8 AM ± 30 minutes, 2 hours post-dose ± 30 minutes, 4 PM ± 30 minutes
Population: Study eye for the Per Protocol population
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Nebivolol Ophthalmic Suspension 1 Percent | Nebivolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Solution 0.5 Percent
Number analyzed (Participants) | 52 | 56 | 55 | 57
mmHg
  Visit 4 - Day 15: number analyzed (Participants) | 51 | 56 | 55 | 57
  Visit 4 - Day 15 | -3.1 (0.44) | -2.2 (0.42) | -5.5 (0.42) | -5.2 (0.41)
  Visit 5 - Day 42: number analyzed (Participants) | 50 | 52 | 55 | 55
  Visit 5 - Day 42 | -3.1 (0.48) | -2.8 (0.47) | -5.4 (0.46) | -5.2 (0.46)
  Visit 6 - Day 84: number analyzed (Participants) | 48 | 49 | 54 | 54
  Visit 6 - Day 84 | -3.5 (0.38) | -3.2 (0.37) | -5.6 (0.36) | -4.9 (0.36)

3. Secondary Outcome: Intraocular Pressure: Change From Baseline at All Time Points at Each Visit
Description: Time-matched change from baseline (Visit 3/Qualification/Baseline) in the 3 daily IOP measurements at Day 15, Day 42 and Day 84
Time Frame: as for outcome 2
Population: Study Eye in the Per Protocol population
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Nebivolol Ophthalmic Suspension 1 Percent | Nebivolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Solution 0.5 Percent
Number analyzed (Participants) | 52 | 56 | 55 | 57
mmHg
  Visit 4 - Day 15 - 8 am: number analyzed (Participants) | 51 | 56 | 55 | 57
  Visit 4 - Day 15 - 8 am | -3.0 (0.49) | -2.5 (0.47) | -6.1 (0.47) | -5.8 (0.47)
  Visit 5 - Day 42 - 8 am: number analyzed (Participants) | 50 | 52 | 55 | 55
  Visit 5 - Day 42 - 8 am | -3.3 (0.52) | -3.4 (0.50) | -5.9 (0.50) | -5.8 (0.49)
  Visit 6 - Day 84 - 8 am: number analyzed (Participants) | 48 | 49 | 54 | 54
  Visit 6 - Day 84 - 8 am | -3.8 (0.48) | -3.7 (0.47) | -6.5 (0.45) | -5.7 (0.45)
  Visit 4 - Day 15 - 10am | -3.2 (0.46) | -2.3 (0.45) | -5.9 (0.45) | -5.5 (0.44)
  Visit 5 - Day 42 - 10 am: number analyzed (Participants) | 49 | 51 | 55 | 55
  Visit 5 - Day 42 - 10 am | -3.3 (0.50) | -3.1 (0.49) | -5.8 (0.48) | -5.2 (0.47)
  Visit 6 - Day 84 - 10 am: number analyzed (Participants) | 47 | 49 | 54 | 54
  Visit 6 - Day 84 - 10 am | -3.4 (0.43) | -3.2 (0.41) | -5.7 (0.40) | -4.9 (0.40)
  Visit 4 - Day 15 - 4 pm | -2.9 (0.43) | -2.4 (0.42) | -4.6 (0.42) | -4.4 (0.41)
  Visit 5 - Day 42 - 4 pm: number analyzed (Participants) | 49 | 50 | 55 | 55
  Visit 5 - Day 42 - 4 pm | -2.7 (0.50) | -2.5 (0.49) | -4.4 (0.48) | -4.5 (0.48)
  Visit 6 - Day 42 - 4 pm: number analyzed (Participants) | 47 | 49 | 54 | 54
  Visit 6 - Day 42 - 4 pm | -3.0 (0.44) | -2.9 (0.43) | -4.7 (0.41) | -4.1 (0.41)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | Nebivolol Ophthalmic Suspension 1 Percent | Nebivolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Suspension 0.5 Percent | Timolol Ophthalmic Solution 0.5 Percent
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/58 | 0/56 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/58 | 0/56 | 0/58
Other Adverse Events (participants affected / at risk) | 7/54 | 6/58 | 7/56 | 6/58
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebivolol Ophthalmic Suspension 1 Percent (N=54) | Nebivolol Ophthalmic Suspension 0.5 Percent (N=58) | Timolol Ophthalmic Suspension 0.5 Percent (N=56) | Timolol Ophthalmic Solution 0.5 Percent (N=58)
Instillation site pain (Eye disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Instillation site reaction (Eye disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Conjunctival hyperemia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Instillation site discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intraocular pressure increased (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT04910100/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04910100/SAP_001.pdf